CLINICAL TRIAL: NCT03431714
Title: Efficacy and Safety of Artesunate-amodiaquine and Dihydroartemisinin-piperaquine for the Treatment of Uncomplicated Falciparum Malaria in Mainland Tanzania
Brief Title: Efficacy and Safety of ASAQ and PD for the Treatment of Uncomplicated Falciparum Malaria in Mainland Tanzania
Acronym: GF-TES-2017
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); World Health Organization (Other)
Responsible Party: Principal Investigator, Dr. Celine Mandara, Researcher, National Institute for Medical Research, Tanzania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIMR-Tanzania
Record Dates: First submitted 2017-12-22; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Uncomplicated Falciparum Malaria
MeSH Terms: interventions — amodiaquine, artesunate drug combination

STUDY DESIGN:
Intervention Model Description: The first group of 88 children were recruited first and given dihydroartemisinin- piperaquine, once the sample size was attained, the second group for artesunate amodiaquine followed and the follow-up for the two groups were running concurrently
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Artesunate amodiaquine tablets containing 25/67.5 mg, 50/135mg and 100/270 mg base of artesunate-amodiaquine were administered according to body weight Dihrdroartemisinin piperaquine tablets containing 160/20mg and 320/40mg base of piperaquine dihydroartemisinin were administered according to body weight
  Interventions: Drug: Artesunate amodiaquine

INTERVENTIONS:
Drug: Artesunate amodiaquine — Drugs were administered under observation of the study nurse for three days
  Other Names: dihydroartemisinin piperaquine

SUMMARY:
The World Health Organization recommends regular surveillance of antimalarial efficacy to monitor the performance of different drugs. The Tanzanian National Malaria Control Programme (NMCP) in collaboration with its partners have been implementing therapeutic efficacy studies (TES) to monitor the performance of different antimalarials in the country. Most of the studies conducted in recent years focused on artemether-lumefantrine which is the first line antimalarial for the treatment of uncomplicated malaria in Mainland Tanzania. However, data on the performance of other artemisinin based combination therapy (ACTs) is urgently needed to support timely review and changes of treatment guidelines in case of drug resistance to current regimen. This study was undertaken in the same NMCP framework to assess the efficacy and safety of alternative ACTs used or with potential use in Tanzania. The study assessed the efficacy and safety of artesunate-amodiaquine (ASAQ) and dihydroartemisinin-piperaquine (DP) for the treatment of uncomplicated malaria in Tanzania. The study was undertaken at two NMCP sentinel sites of Kibaha and Ujiji from July to December 2017.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 months to 10 years.
* mono-infection with P. falciparum detected by microscopy;
* parasitaemia of 250 - 200,000/μl asexual forms;
* presence of axillary temperature ≥37.5 °C or history of fever during the past 24 hours
* ability to swallow oral medication;
* ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule; and
* Informed consent from the parents or guardians of children.

Exclusion Criteria:

* mRDT negative
* presence of general danger signs in children aged 6 months to 10 years or signs of severe falciparum malaria according to the definitions of WHO (Appendix 1);
* weight under 5 Kg
* mixed or mono-infection with another Plasmodium species detected by microscopy;
* presence of severe malnutrition (defined as a child who has symmetrical oedema involving at least the feet or has a mid-upper arm circumference < 110 mm in children ≤ 59 months; or BMI of <16 in children aged 5 years and above)
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* regular medication, which may interfere with antimalarial pharmacokinetics;
* history of hypersensitivity reactions or contraindications to any of the medicine(s) being tested or used as alternative treatment(s);

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Adequate clinical response | 28 days
  Proportions of patients with 100% cure before PCR correction

SECONDARY OUTCOMES:
PCR corrected responses | one months after study completion
  Proportions of patients with 100% cure after PCR correction

CONTACTS AND LOCATIONS:
Overall Officials: Deus S Ishengoma, PhD, Principal Investigator — National Institute for Medical Research
Locations (1):
- National Institute for Medical Research, Tanga, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mandara CI, Francis F, Chiduo MG, Ngasala B, Mandike R, Mkude S, Chacky F, Molteni F, Njau R, Mohamed A, Warsame M, Ishengoma DS. High cure rates and tolerability of artesunate-amodiaquine and dihydroartemisinin-piperaquine for the treatment of uncomplicated falciparum malaria in Kibaha and Kigoma, Tanzania. Malar J. 2019 Mar 25;18(1):99. doi: 10.1186/s12936-019-2740-z. PMID 30909922